CLINICAL TRIAL: NCT01821560
Title: Baclofen Effects on Brain and Behavior in Cigarette Smokers
Brief Title: Baclofen Effects in Cigarette Smokers
Acronym: BAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 817101; R01DA030394-01A1 (NIH); PA Depart of Health (Other Grant/Funding Number: CURE (Commonwealth Universal Research Enhancement) Program)
Record Dates: First submitted 2013-03-21; First posted 2013-04-01 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Nicotine Dependence
Keywords: Nicotine Addiction; fMRI; Baclofen
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo-treated subjects will follow the identical schedule as Baclofen subjects.
  Interventions: Drug: placebo
- Baclofen (Active Comparator): Baclofen will be dispensed in pill form. Baclofen will be prescribed at 20 mg 4 times per day. Each baclofen pill will be 10 mg. Thus, 2 pills will be taken at each scheduled dose for a total of 8 pills a day over a period of 8 weeks. In this way, the titration schedule, taper and potential dose reductions can be managed.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen
  Other Names: Kemstro; Lioresal; Liofen; Gablofen; Beklo
  Arms: Baclofen
Drug: placebo
  Arms: Sugar pill

SUMMARY:
The proposed project will utilize perfusion functional magnetic resonance imaging (fMRI), a functional candidate gene association approach (of dopaminergic addictions-targeted polymorphisms), and the dopamine-modulating and gamma-aminobutyric acid (GABA) B receptor agonist, baclofen, to examine the brain and behavioral responses in smokers to appetitive smoking reminders (cues that motivate continued smoking and relapse). These studies will provide a means to identify an appetitive cue-sensitive pharmacologic-responsive endophenotype. Once brain/behavioral/genetic endophenotypes can be determined prior to treatment, smoking cessation treatments can be structured to meet individual needs, which will significantly improve treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy, as determined by a comprehensive physical examination and approval of the study physician males or females who smoke cigarettes, ages 18-60.
* Smoke ≥ 6 cigarettes per day for at least 6 months prior to study start date.
* Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of child bearing potential but practicing a medically acceptable method of birth control. Examples of medically acceptable methods for this protocol include barrier (diaphragm or condom) with spermicide, an intrauterine device (IUD), the Nuvaring, oral contraceptives, levonorgestrel implant, hormonal injection or complete abstinence.
* Provide voluntary informed consent.
* Must be able to read. [Subjects are required to be able to read because there are several self-administered measures that they must read, understand and provide written answers.]
* Intelligence quotient of ≥ 80.

Exclusion Criteria:

* History of head trauma or injury causing loss of consciousness, lasting more than five (5) minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI.
* Current Diagnostic and Statistical Manual-IV (DSM-IV) Axis I diagnoses other than nicotine dependence.
* Presence of magnetically active irremovable prosthetics, plates, pins, permanent retainer, bullets, etc. (unless a radiologist confirms that it's presence is unproblematic). An x-ray may be obtained to determine eligibility given the possibility of a foreign body.
* History of psychosis.
* Claustrophobia or other medical condition preventing subject from lying in the MRI for approximately one (1) hour.
* Current diagnosis of or treatment within the last 3 months for alcohol dependence.
* Current use of any smoking cessation treatments such as Zyban, Chantix, Wellbutrin, patch, gum, inhaler, electronic cigarettes, herbal preparations.
* Vision problems that cannot be corrected with glasses.
* Weight exceeding 300 pounds [Imaging data acquisition is impaired with high weight individuals].
* History of stroke.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa R Franklin, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruitment between March 2013-March 2017 via word of mouth, flyers, an online study database managed by the University of Pennsylvania, and also social media advertisements (Facebook).
Pre-assignment Details: Prior to study group assignments, all participants must first provide informed consent and then are found to be eligible to participate in the study after completing the screening process. The screening process included a full physical and psychological evaluation to ensure all participants are both physically and mentally healthy enough.
Groups:
- Sugar Pill: Placebo-treated subjects will follow the identical schedule as Baclofen subjects.
  placebo
- Baclofen: Baclofen will be dispensed in pill form. Baclofen will be prescribed at 20 mg 4 times per day. Each baclofen pill will be 10 mg. Thus, 2 pills will be taken at each scheduled dose for a total of 8 pills a day over a period of 8 weeks. In this way, the titration schedule, taper and potential dose reductions can be managed.
  Baclofen
Period: Overall Study
Arm/Group | Sugar Pill | Baclofen
Started | 22 | 22
Completed | 16 | 15
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Baclofen | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (12.1) | 38.9 (12.0) | 39.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 14 | 12 | 26
  Race: White Non-Hispanic | 3 | 5 | 8
  Race: Asian | 2 | 2 | 4
  Race: Mixed Race | 0 | 2 | 2
  Race: White Hispanic | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Smoked Per Day
Description: Cigarettes per day at Scan Day 2; Baclofen group vs. placebo group
Time Frame: 3 weeks (Scan Day 1, week1- Scan Day 2, week 4)
Measure: Mean (Standard Error); unit: Cigarettes per day
Arm/Group | Sugar Pill | Baclofen
Number analyzed (Participants) | 22 | 22
Cigarettes per day
  Scan Day 1 | 14.19 (1.01) | 14.23 (1.20)
  Scan Day 2 | 7.67 (1.05) | 7.76 (1.10)

ADVERSE EVENTS:
Time Frame: Collected over a 5 year period
Arm/Group | Sugar Pill | Baclofen
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 17/22 | 16/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=22) | Baclofen (N=22)
Drowsiness (Nervous system disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 4 | 2
Dizzy/Lightheadedness (Nervous system disorders) | 1 | 5
Insomnia (Nervous system disorders) | 1 | 2
Cognitive Changes (Nervous system disorders) | 2 | 4 — vivid Dreams, nightmares, mental fogginess
Affective Changes (Psychiatric disorders) | 0 | 4 — irritability, mood swings
Elevated Blood Pressure (Vascular disorders) | 1 | 3
Digestive (Gastrointestinal disorders) | 4 | 4 — gas, heartburn, increased appetite, decreased appetite, bowel changes, diarrhea, stomach pain
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 2 — muscle weakness

LIMITATIONS AND CAVEATS:
The goals of the study were to identify mechanisms of baclofen's effects on smoking cue reactivity. Using other mechanisms we provided a treatment arm. Sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT01821560/Prot_SAP_000.pdf